CLINICAL TRIAL: NCT06145035
Title: University of Louisville - 18642 / CATO Study, Single or Repeated Intravenous Administration of umbiliCAl Cord Mesenchymal sTrOmal Cells in Ischemic Cardiomyopathy
Brief Title: Single or Repeated Intravenous Administration of umbiliCAl Cord Mesenchymal sTrOmal Cells in Ischemic Cardiomyopathy
Acronym: CATO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roberto Bolli (Other)
Collaborators: University of Miami (Other); University of Texas (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Roberto Bolli, Endowed Chair, M.D., University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23.0712; 1369707 (Other Grant/Funding Number: United States Department of Defence)
Record Dates: First submitted 2023-11-01; First posted 2023-11-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Heart Disease
Keywords: ischemic cardiopathy; UC-MSCs
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled,
Who Masked: Participant, Investigator
Masking Description: As a double-blind study, bias control will be achieved by maintaining the blind on treatment group assignments. The master randomization lists containing the treatment assignments will be protected in secure, controlled access drives/folders and will not be released to any blinded study personnel prior to final database lock. A centralized Core laboratory will be used for MRI analyses to maintain the blind across the study team.
  The designated cell processing technicians will prepare the investigational product for infusion. The investigational agent infusions will be prepared in identical infusion bags and labeled with the identical investigational drug labels as to preserve the blind. The designated technicians in the ISCI Cell Processing Laboratory (CPL) or designee will be responsible for maintaining the investigational product records including randomized treatment assignments by subject identification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): Four doses of vehicle (Plasma-Lyte A supplemented with 1% HSA) will be given 2 months apart. Each dose will be infused IV at a rate of 2 ml/min for a total of 60 ml over 30 minutes.
  Interventions: Biological: umbilical cord-derived mesenchymal stromal cells (UC-MSCs)
- single-dose group (Experimental): One dose of UC-MSCs (100 x 106 cells) will be infused IV at a rate of 2 ml/min for a total of 60 ml over 30 minutes (3.3 million cells/ml/min). This will be followed by three IV infusions of placebo (same volume and rate) 2, 4, and 6 months later.
  Interventions: Biological: umbilical cord-derived mesenchymal stromal cells (UC-MSCs)
- repeated-dose group (Experimental): Four doses of UC-MSCs (100 x 106 cells each) will be given 2 months apart. Each dose will be infused IV at a rate of 2 ml/min for a total of 60 ml over 30 minutes (3.3 million cells/ml/min).
  Interventions: Biological: umbilical cord-derived mesenchymal stromal cells (UC-MSCs)

INTERVENTIONS:
Biological: umbilical cord-derived mesenchymal stromal cells (UC-MSCs) — The study product will consist of 100 million UC-MSCs suspended in a final volume of 60 ml given at a rate of 3.3 million cells/min. The product will be infused into vein via intravenous line placed in the arm.

SUMMARY:
This is a Phase IIA, randomized, double blind, placebo controlled, multicenter study designed to assess the safety, feasibility, and efficacy of umbilical cord derived mesenchymal stromal cells (UC MSCs), administered intravenously (IV) as a single dose or repeated doses, in patients with ischemic cardiomyopathy (ICM).

DETAILED DESCRIPTION:
This is a Phase IIA, randomized, double blind, placebo controlled, multicenter study designed to assess the safety, feasibility, and efficacy of umbilical cord derived mesenchymal stromal cells (UC MSCs), administered intravenously (IV) as a single dose or repeated doses, in patients with ischemic cardiomyopathy (ICM) (see summary in Figure 1).

A total of 60 participants will be assigned in a random fashion to three groups on a 1:1:1 basis: control, single dose, and repeated doses. All patients will receive four study product infusions (SPIs) 2 months apart. SPIs (performed in a double blind fashion) will consist of either UC MSCs or placebo (based on randomization), infused by the IV route. Patients in the control group will receive four doses of placebo. Patients in the single dose group will receive one dose of UC MSCs followed by three doses of placebo. Patients in the repeated dose group will receive four doses of UC MSCs. A dose of UC MSCs will consist of 100 million cells suspended in 60 mL, infused at a rate of 2 mL/min. A dose of placebo will consist of an equivalent volume of Plasma Lyte A supplemented with 1% human serum albumin (HSA). After each SPI, patients will be monitored for a minimum of 2 hours and then examined at 1 week and 2 months. After the fourth SPI, patients will be followed for 6 months to complete all safety and efficacy assessments.

The UC MSCs will be derived from UC tissue obtained from a healthy pregnant woman at the time of caesarean delivery. The cells will be manufactured at the Interdisciplinary Stem Cell Institute at the University of Miami, Miller School of Medicine and then shipped to the Site for administration.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 21 and ≤ 85 years of age.
2. Have documented CAD (> 70% lesion in at least 1 epicardial vessel) with evidence of myocardial injury, LV dysfunction, and clinical evidence of HF.
3. Have a "detectable" area of myocardial injury defined as ≥ 5% LV involvement (infarct volume) and any subendocardial involvement by MRI.
4. Have an EF ≤ 40% by MRI.
5. Be receiving guideline driven medical therapy for HF (beta blockers, diuretics, ACE inhibitors or ARBs, or ARNIs, aldosterone antagonists, hydralazine isosorbide, sodium-glucose transporter 2 inhibitors) ) at stable, maximally tolerated doses for ≥ 1 month prior to consent. "Stable" is defined as stable dose with no changes for 30 days after last dose adjustment. For beta blockade "stable" is defined as no greater than a 50% reduction in dose or no more than a 100% increase in dose.
6. Have NYHA class I, II or III symptoms of HF (see Appendix A)
7. If a female of childbearing potential, be willing to use one form of birth control for the duration of the study and undergo a serum pregnancy test at baseline and within 36 hours prior to infusion

Exclusion Criteria:

1. Indication for standard of care surgery (including valve surgery, placement of left ventricular assist device, or imminent heart transplantation), coronary artery bypass grafting (CABG) procedure, and/or percutaneous coronary intervention (PCI) for the treatment of ischemic and/or valvular heart disease. Subjects who require or undergo PCI should undergo these procedures a minimum of 3 months in advance of randomization. Subjects who require or undergo CABG should undergo these procedures a minimum of 3 months in advance of randomization. In addition, subjects who develop a need for revascularization following enrollment should undergo revascularization without delay. Indication for imminent heart transplantation is defined as a high likelihood of transplant prior to collection of the 12 month study endpoint. Candidates cannot be UNOS 1A or 1B, and they must have documented a low probability of being transplanted.
2. Severe valvular (any valve) insufficiency and/or regurgitation within 12 months of consent
3. History of ischemic or hemorrhagic stroke within 90 days of consent
4. Presence of a pacemaker and/or implantable cardiac device (ICD) generator with any of the following limitations/conditions:

   * manufactured before the year 2000
   * leads implanted < 6 weeks prior to consent
   * non transvenous epicardial or abandoned leads
   * subcutaneous ICDs (if not MRI compatible)
   * leadless pacemakers
   * any other condition that, in the judgment of device trained staff, would deem an MRI contraindicated
5. Pacemaker dependence with an ICD (Note: pacemaker dependent candidates without an ICD are not excluded)
6. A cardiac resynchronization therapy (CRT) device implanted less than 3 months prior to consent.
7. Other MRI contraindications (e.g. patient body habitus incompatible with MRI)
8. An appropriate ICD firing or anti tachycardia pacing (ATP) for ventricular fibrillation or ventricular tachycardia within 30 days of consent
9. Ventricular tachycardia ≥ 20 consecutive beats without an ICD within 3 months of consent, or symptomatic Mobitz II or higher degree atrioventricular block without a functioning pacemaker within 3 months of consent
10. Evidence of active myocarditis
11. Baseline glomerular filtration rate (eGFR) < 35 ml/min/1.73m2
12. Blood glucose levels (HbA1c) >10%
13. Hematologic abnormality evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet count < 100,000/ul
14. Liver dysfunction evidenced by enzymes (AST and ALT) ˃ 3 times the ULN.
15. HIV and/or active HBV or HCV
16. Known history of anaphylactic reaction to penicillin or streptomycin
17. Received gene or cell based therapy from any source within the previous 12 months.
18. History of malignancy within 2 years (i.e., subjects with prior malignancy must be disease free for 2 years), excluding basal cell carcinoma and cervical carcinoma in situ which have been definitively treated.
19. Condition that limits lifespan to < 1 year
20. History of drug abuse (illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 12 months.
21. Participation in an investigational therapeutic or device trial within 30 days of consent
22. Cognitive or language barriers that prohibit obtaining informed consent or any study elements
23. Pregnancy or lactation or plans to become pregnant in the next 12 months.
24. Any other condition that, in the judgment of the Investigator or Sponsor, would impair enrollment, study product administration, or follow up.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
change in LVEF (D LVEF) between baseline (M0) and 12 months after the first study product infusion (SPI) (M12) | Baseline, 12 months
  Change in left ventricular ejection fraction as assessed via cardiac MRI. Units: %

SECONDARY OUTCOMES:
Change in LV end-systolic volume index (ESVI) | Baseline, 12 months
  Change in left ventricular end systolic index (LVESVI) as assessed via cardiac MRI.
  Units: ml/m2
Change in LV end-diastolic volume index (EDVI) | Baseline, 12 months
  Change in left ventricular end diastolic index (LVEDVI) as assessed via cardiac MRI.
  Units: ml/m2
Change in LV end-diastolic wall thickness | Baseline, 12 months
  Change in LV end-diastolic wall thickness as assessed via cardiac MRI. Units: mm
Change in LV wall thickening | Baseline, 12 months
  Change in LV wall thickening as assessed via cardiac MRI. Units: mm
Change in LV sphericity index | Baseline, 12 months
  Change in LV sphericity index as assessed via cardiac MRI. Units: Index score Sphericity index is the ratio of the long and short axis measurements of the left ventricle.
Change in global and regional strain (tagged MRI): global and 16-segment values for peak circumferential strain, global and segmental longitudinal strain | Baseline, 12 months
  Change in global and regional strain as assessed via cardiac MRI. Units: %
Change in scar mass (in grams) | Baseline, 12 months
  Change in scar mass (in grams) as assessed via delayed gadolinium enhancement MRI.
  Units: grams
Change in scar mass (as %LV) | Baseline, 12 months
  Change in scar mass (as %LV) as assessed via delayed gadolinium enhancement MRI.
  Units: %
Change in VO2 max (treadmill test) | Baseline, month 8, month 12
  Change in maximal oxygen consumption (peak VO2) as assessed via treadmill. Units: mL/kg/min
Change in exercise tolerance (six-minute walk test) | Baseline, month 8, month 12
  Change in exercise tolerance as assessed as the distance covered via the six-minute walk test.
  Units: meters
Change in New York Heart Association class | Baseline, month 2,4,6,8, & 12
  NYHA Classifications of heart failure are as follows: Class I (no limitations); Class II (mild symptoms); Class III (marked limitations); Class IV (Severe limitations).
  Units: score on a scale
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Baseline, month 6, month 12
  KCCQ is a 12-item questionnaire in which scores are scaled from 0 to 100 and summarized in ranges to represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
  Units: score on a scale
Change in Endothelial Progenitor Cell [EPC]-colony forming unit [EPC-CFU] assay | Baseline, month 2, 8, & 12
  Change in endothelial function will be reported as the change in Endothelial Progenitor Cell Colony Forming Unit (EPC-CFU) assessed via blood sample assay.
  Units: CFUs/well
Change in branchial artery flow-mediated dilation [FMD] [diameter percent change]). | Baseline, month 2, 8, & 12
  Change in branchial artery flow-mediated dilation will be reported as the percent change in flow mediated diameter assessed via flow mediated dilation (FMD).
  Units: %
Major adverse cardiac events (MACE) | Month 12
  Number of participants with adjudicated events including death, hospitalization for worsening HF, and exacerbation of HF requiring visit to the Emergency Department and/or IV therapy but not requiring hospitalization.
  Units: number of participants who have an incidence of MACE in each group
Cumulative days alive and out of hospital for HF | Month 12
  Days alive and out of hospital during the study evaluation period. Units: days
Biomarkers: Change in NT-proBNP | Day 0, Month 2, 4, 6, 8, & 12
  Change in NT-proBNP as assessed via blood draw. Units: pg/ml
Biomarkers: hs-CRP | Day 0, Week 1, Month 2, 4, 6, 8, & 12
  Blood level of hs-CRP as assessed via blood draw. Units: mg/ml

OTHER OUTCOMES:
Serious adverse events | 2 hrs, 6 hrs, Months 2 & 6
  Number of patients experiencing significant adjudicated clinical events including myocardial infarction (MI), stroke, pulmonary embolism, implantable cardioverter-defibrillator (ICD) firing for ventricular fibrillation/tachycardia, ventricular tachycardia (sustained and non-sustained), or hospitalization related to intravenous infusion of UC-MSCs.
  Units: number of participants who have an incidence of SAE in each group

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bolli, MD, Principal Investigator — University of Louisville School of Medicine
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Louisville School of Medicine, Institute of Molecular Cardiology, Louisville, Kentucky
  - The Texas Heart Institute Houston Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolli R, Tang XL, Hare JM, Mitrani RD, Perin EC, Lima JA, Hurwitz BE, Kalra D, Singh G, Saltzman RG, Caceres LV, Nettina A, Lee YS, Bacallao K, Grant E, Khan A. Design and rationale of CATO, a Phase IIA, randomized, double-blind, placebo-controlled study of single or repeated intravenous administration of umbilical cord-derived mesenchymal stromal cells in ischemic cardiomyopathy. Am Heart J. 2025 Dec 13;294:107328. doi: 10.1016/j.ahj.2025.107328. Online ahead of print. PMID 41397478
- [Derived] Tang XL, Wysoczynski M, Gumpert AM, Solanki M, Li Y, Wu WJ, Zheng S, Ruble H, Li H, Stowers H, Zheng S, Ou Q, Tanveer N, Slezak J, Kalra DK, Bolli R. Intravenous infusions of mesenchymal stromal cells have cumulative beneficial effects in a porcine model of chronic ischaemic cardiomyopathy. Cardiovasc Res. 2024 Dec 4;120(15):1939-1952. doi: 10.1093/cvr/cvae173. PMID 39163570